CLINICAL TRIAL: NCT06093204
Title: The Potential Role of Compounds Derived From Ultra-processed Foods in Pathogenesis of Eosinophilic Esophagitis
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, MD,PhD,Prof., Federico II University
Other Study IDs: 00014834
Record Dates: First submitted 2023-07-26; First posted 2023-10-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Esophagitis, Eosinophilic
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with eosinophilic esophagitis: Patients with a sure diagnosis of eosinophilic esophagitis
  Interventions: Other: Dietary evaluation
- Sex and age matched healthy controls: Matched healthy controls for age and gender, without eosinophilic esophagitis
  Interventions: Other: Dietary evaluation

INTERVENTIONS:
Other: Dietary evaluation — Comparative evaluation of the dietary consumption of ultraprocessed foods and ultraprocessed foods-derived compounds

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic antigen-mediated inflammatory disease of the esophagus that affects both children and adults. The incidence and prevalence of EoE is rapidly increasing in Western countries with an estimated incidence of 6.6 per 100,000 person-years (95% CI, 3-11.7) in children and 7.7 per 100,000 person-years (95% CI, 1.8-17.8) in adults. Clinically, it is characterized by various symptoms related to esophageal dysfunction, including vomiting, regurgitation, feeding difficulties, epigastric heartburn, dysphagia, or food bolus impaction, and may cause growth retardation. Diagnosis is made on the basis of clinical symptoms and histological evidence of eosinophilic infiltration of the esophagus (at least 15 eosinophils/high power microscope field (eos /hpf), excluding other etiologies of esophageal eosinophilia (gastroesophageal reflux disease, infectious esophagitis, achalasia, celiac disease and Crohn's disease, connective tissue disorders, gra ft versus host disease, drug hypersensitivity and hypereosinophilic syndromes). EoE is primarily characterized by a T helper 2 type inflammation, but the pathogenesis and the immunopathological mechanisms underlying the pathology are not yet fully understood. Recent evidence suggests that in genetically predisposed individuals, interaction with environmental factors (e.g., dietary lifestyle) may play a role in activating several inflammatory pathways and cause EoE.

Ultra-processed foods (UPFs) are food and beverage products resulting from industrial formulations, ready for consumption, typically obtained with five or more ingredients from different manufacturing processes (cooking methods, addition of additives such as stabilizers or preservatives). During the last decade, the consumption of the latter has increased significantly among the pediatric population to represent 30% of the daily caloric intake of an average child in Europe and America. Recent evidences show that UPFs favor the onset of chronic non-communicable diseases through the activation of different inflammatory pathways.

The components mostly represented in UPFs are the advanced glycation end products (AGEs), a heterogeneous group of highly oxidizing compounds that are formed through non-enzymatic reactions (Maillard reaction) between reduced sugars and free amino groups of proteins, lipids, or nucleic acids.

Evidence demonstrates that dietary AGEs are absorbed and contribute significantly to the total concentration of AGEs in the body. AGEs induce oxidative stress and inflammation, leading to structural and functional protein alterations, cellular apoptosis and multi-tissue/organ damage. These mechanisms are mediated at least in part by interactions with their cell-surface receptor for advanced glycation end-products (RAGE).

The AGEs-RAGE interaction modulates the immune response. AGEs are able to activate le mast cells, to stimulate the release of histamine and to induce a chronic inflammatory state that promotes a T helper 2 type response.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* age between 3-65 years
* sure diagnosis of eosinophilic esophagitis
* age- and sex-matched healthy controls
* parents/tutor written informed consent.

Exclusion Criteria:

* lack of written informed consent;
* non-Caucasian ethnicity
* age at enrollment < 3 or >65 years
* simultaneous presence of other chronic diseases: eosinophilic gastroenteritis, eosinophilic colitis, achalasia, GERD, hypereosinophilia syndrome, IBD, fungal or viral infections, connective tissue disorders, autoimmune diseases, vasculitis, bullous dermatosis with oesophageal involvement (pemphigus), drug hypersensitivity reactions, drug-induced oesophagitis, graft vs host disease, monogenic disorders (Marfan syndrome type 2, HIES, PTEN).
* presence of tattoos, scars, moles or particular lesions on both forearms

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients both sexes, aged between 3-65 years with diagnosis of eosinophilic esophagitis and age- and sex-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Comparative evaluation of the dietary consumption of Ultraprocessed Foods | At enrollment
  A 7-day food diary to evaluate the dietary intake of ultraprocessed foods.

SECONDARY OUTCOMES:
Intake of dietary Advanced Glycation End-products | At enrollment
  A 7-day food diary to evaluate the dietary intake of the detrimental compounds of ultraprocessed foods, the advanced glycation end-products.
Skin Advanced Gycation End-products accumulation level | At enrollment
  AGEs reader to evaluate the skin Advanced Gycation End-products accumulation level. Skin AGEs levels will be calculated as the ratio between the emission light and reflected excitation light, multiplied by 100 and expressed in arbitrary units (AU).
Advanced Glycation End-Products receptor (RAGE) expression in peripheral blood mononuclear cells (PBMCs) | At enrollment
  ELISA test.
Advanced Glycation End-Products receptor (RAGE) expression in plasma | At enrollment
  ELISA test
Advanced Glycation End-Products receptor (RAGE) expression in peripheral blood mononuclear cells (PBMCs) | At enrollment
  flow cytometry
Disease severity | At 3 months, at 6 months
  Pediatric Eosinophilic Esophagitis Symptom Scores (PEES Score)
Disease severity | At 3 months, at 6 months
  Eosinophilic Esophagitis Endoscopic Reference Score (EREFS Score)
Treatment response | At 3 months, at 6 months
  Drug used for inducing eosinophilic esophagitis remission defined as <15 eosinophils per high-power field (eos/hpf)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No